CLINICAL TRIAL: NCT00502255
Title: Telemonitoring in Patients With Heart Failure
Acronym: TEHAF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Josiane Boyne, RN,MA, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 072036
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Heart Failure, Congestive
Keywords: Telemonitoring; Cost-effectiveness; Heart failure; Case management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telemonitoring (Experimental): Health Buddy in patients home situation
  Interventions: Device: Health Buddy system
- usual care (Experimental): patients receive care as usual
  Interventions: Device: Telemonitoring in patients with heart failure

INTERVENTIONS:
Device: Health Buddy system — Patients are followed on distance by the Health Buddy system.
  Other Names: TEHAF study; Therapy compliance in patients with heart failure; Cost effectiveness
  Arms: telemonitoring
Device: Telemonitoring in patients with heart failure — Health Buddy in patients home situation.
  Other Names: TEHAf study
  Arms: usual care

SUMMARY:
The purpose of this study is to investigate if telemonitoring results in a decrease in hospital admissions, with equal quality of care defined as mortality, quality of life and unplanned visits with caregivers. Telemonitoring is expected to be more cost-effective than usual care in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Patients with heart failure NYHA classification II-III-IV
* Patient experienced a period of fluid retention
* Patient is treated by a cardiologist
* Patient is followed-up by a heart failure nurse
* Adequate knowledge of the Dutch language
* Patient has an active telephone connection, preferably analogue
* Patient is mental competent
* Patient has the disposal of a balance

Exclusion Criteria:

* Patients suffering from COPD, Gold classification 3 or 4
* Patient is a dialysis patient
* Patient has a visual restriction to read the dialogues on the Health Buddy
* Patient is hard of hearing or deaf
* Patient suffers from a lethal sickness with a prognosis < 1 year
* Patient participates in another trial
* Patient needs a hospital admission on short time, i.e., < 3 months
* Patient used the Health Buddy in an earlier stage
* Patient is an illiterate person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2007-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To what extent does the use of Health Buddy result in a decrease in hospital admissions? | one year
To what extent is Health Buddy® more cost-effective than usual care? | one year
To what extent will the amount of planned contacts decrease without an increase of unplanned contacts? | one year

SECONDARY OUTCOMES:
What is the effect of Health Buddy® in patients with heart failure in regard to drug consumption and therapy compliance and level of knowledge, and quality of life? | one year
To what extent is it - based on patients' characteristics - possible to identify patient with benefits? | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hubertus J Vrijhoef, Dr, Study Chair — University Maastricht
Locations (3):
- Netherlands (3):
  - Atrium Medische Centrum, Heerlen, Limburg
  - Maastricht University Hospital, Maastricht, Limburg
  - Orbis Medische en Zorgconcern, Sittard, Limburg

REFERENCES:
- [Derived] Boyne JJ, Vrijhoef HJ, Crijns HJ, De Weerd G, Kragten J, Gorgels AP; TEHAF investigators. Tailored telemonitoring in patients with heart failure: results of a multicentre randomized controlled trial. Eur J Heart Fail. 2012 Jul;14(7):791-801. doi: 10.1093/eurjhf/hfs058. Epub 2012 May 15. PMID 22588319
- [Derived] Boyne JJ, Vrijhoef HJ, Wit Rd, Gorgels AP. Telemonitoring in patients with heart failure, the TEHAF study: Study protocol of an ongoing prospective randomised trial. Int J Nurs Stud. 2011 Jan;48(1):94-9. doi: 10.1016/j.ijnurstu.2010.05.017. Epub 2010 Jul 7. PMID 20615505